CLINICAL TRIAL: NCT01285518
Title: A Phase 1, Placebo-controlled, Randomized Study To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Following Single, Escalating Intravenous Doses Of Pf-05231023 In Adult Subjects With Type 2 Diabetes
Brief Title: Safety And Tolerability Of Escalating Intravenous Doses Of PF-05231023 In Adult Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2901001
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; intravenous; single dose
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — PF-05231023

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Drug: PF-05231023
- Placebo (Placebo Comparator): 0.9% w/v sodium chloride injection, USP
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-05231023 — 0.5 mg QD IV x 1 day
  Arms: Treatment
Drug: PF-05231023 — 1.5 mg QD IV x 1 day
  Arms: Treatment
Drug: PF-05231023 — 5 mg QD IV x 1 day
  Arms: Treatment
Drug: PF-05231023 — 15 mg QD IV x 1 day
  Arms: Treatment
Drug: PF-05231023 — 50 mg QD IV x 1 day
  Arms: Treatment
Drug: PF-05231023 — 100 mg QD IV x 1 day
  Arms: Treatment
Drug: PF-05231023 — 200 mg QD IV x 1 day
  Arms: Treatment
Other: Placebo — 0.9% w/v sodium chloride injection, USP QD IVx 1 day
  Arms: Placebo

SUMMARY:
This is a trial in subjects with Type 2 diabetes mellitus to study the safety, tolerability and pharmacokinetics and pharmacodynamics of single escalating doses of PF-05231023.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 30 and 65 years, inclusive, with a historical diagnosis of type 2 diabetes mellitus, diagnosed according to the American Diabetes Association guidelines.
* Body Mass Index (BMI) of 25 to 35.5 kg/m2, and a total body weight >50 kg (110 lbs).
* HbA1c >7% and not to exceed 10.5%.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Diagnosis of Type 1 diabetes mellitus
* Evidence of diabetic complications with significant end organ damage.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Profil Institute for Clinical Research, Inc., Chula Vista, California
  - Comprehensive Phase One (A Division of Comprehensive NeuroScience, Inc.), Fort Meyers, Florida
  - Elite Research Institute, Miami, Florida
  - Comprehensive Phase One (A Division of Comprehensive NeuroScience, Inc.), Miramar, Florida
  - Cetero Research, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2901001&StudyName=Safety%20And%20Tolerability%20Of%20Escalating%20Intravenous%20Doses%20Of%20PF-05231023%20In%20Adult%20Subjects%20With%20Type%202%20Diabetes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a historical diagnosis of type 2 diabetes mellitus (T2DM), diagnosed according to the American Diabetes Association (ADA) guidelines and those with well-controlled diabetes were recruited in the study.
Pre-assignment Details: Dose of PF-05231023 was escalated based on sponsor's and investigator's discretion, depending upon safety, tolerability and pharmacokinetic profile of PF-05231023.
Groups:
- PF-05231023 0.5 mg: Single dose of PF-05231023 0.5 milligram (mg) intravenous bolus injection on Day 1.
- PF-05231023 1.5 mg: Single dose of PF-05231023 1.5 mg, intravenous bolus injection on Day 1.
- PF-05231023 5 mg: Single dose of PF-05231023 5 mg intravenous infusion over approximately 1 hour on Day 1.
- PF-05231023 15 mg: Single dose of PF-05231023 15 mg intravenous infusion over approximately 1 hour on Day 1.
- PF-05231023 50 mg: Single dose of PF-05231023 50 mg intravenous infusion over approximately 1 hour on Day 1.
- PF-05231023 100 mg: Single dose of PF-05231023 100 mg intravenous infusion over approximately 1 hour on Day 1.
- PF-05231023 200 mg: Single dose of PF-05231023 200 mg intravenous infusion over approximately 1 hour on Day 1.
- Placebo: Single dose of placebo matched to either intravenous bolus injection or intravenous infusion over approximately 1 hour on Day 1.
Period: Overall Study
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Started | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
Completed | 10 | 10 | 10 | 10 | 10 | 9 | 10 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (4.1) | 58.4 (3.9) | 53.8 (7.2) | 53.3 (8.2) | 54.5 (8.6) | 55.2 (7.3) | 57.2 (5.7) | 52.9 (6.8) | 55.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 2 | 3 | 2 | 3 | 5 | 24
  Male | 6 | 7 | 8 | 8 | 7 | 8 | 7 | 9 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: Physical examination included assessment of height, weight, blood pressure and pulse rate. Criteria for abnormal physical findings was based on investigator's discretion and were reported as adverse event (AE), as planned.
Time Frame: Day -1 up to Day 22
Population: Data was not collected since this outcome measure was not analyzed as per Sponsor's discretion.
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 22 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 up to Day 22
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
participants
  AEs | 4 | 3 | 3 | 2 | 7 | 2 | 8 | 5
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Abnormal Laboratory Values
Description: Criteria for laboratory tests abnormalities included: hemoglobin, hematocrit and red blood cells (RBCs)(less than [<] 0.8*lower limit of normal[LLN]); leucocytes (<0.6/greater than [>]1.5*upper limit of normal [ULN]); platelets (<0.5*LLN/>1.75*ULN); neutrophils, lymphocytes (<0.8*LLN/>1.2*ULN); eosinophils, basophils, monocytes (>1.2*ULN); total bilirubin, direct bilirubin, indirect bilirubin (>1.5*ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (>3*ULN), total protein, albumin (<0.8*LLN/>1.2*ULN); creatinine, urea (>1.3*ULN); glucose (<0.6*LLN/>1.5*ULN); uric acid (>1.2*ULN); sodium, potassium, chloride, calcium, bicarbonate (<0.9*LLN/>1.1*ULN); urine RBCs, urine white blood cells (WBCs) (> or equal[=]20 high-powered field), urine bacteria >20 high-powered field. Total number of participants with any laboratory abnormalities was reported.
Time Frame: Day -1 up to Day 15
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
participants | 9 | 9 | 9 | 8 | 10 | 6 | 6 | 14

4. Primary Outcome: Number of Participants With Vital Signs Abnormalities
Description: Criteria for vital signs abnormalities: supine systolic blood pressure (SBP) <90 millimeter of mercury (mmHg), supine diastolic BP (DBP) <50 mmHg, supine pulse rate <40 beats per minute (bpm). Maximum increase or decrease from baseline in supine SBP >=30 mmHg and maximum increase or decrease from baseline in supine DBP >=20 mmHg.
Time Frame: Day 1 up to Day 15
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
participants
  Supine SBP <90 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Supine DBP <50 mmHg | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine pulse rate <40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine pulse rate >120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Supine SBP: Maximum increase >=30 mmHg | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 0
  Supine DBP: Maximum increase >=20 mmHg | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Supine SBP: Maximum decrease >=30 mmHg | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 1
  Supine DBP: Maximum decrease >=20 mmHg | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1

5. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Criteria for potential clinical concern in ECG parameters: maximum PR interval of greater than or equal to (>=) 300 milliseconds (msec), maximum QRS interval >=140 msec, maximum QTCF interval (Fridericia's Correction) of 450 to <480 msec, 480 to <500 msec and >=500 msec, maximum increase of >=25 percent (%) for baseline value of >200 msec for PR interval and maximum increase of >=50% for baseline value of less than or equal to (<=) 200 msec for QRS interval, maximum increase from baseline of >=30 msec to <60 msec and maximum increase from baseline of >60 msec in QTCF interval (Fridericia's Correction).
Time Frame: Screening up to Day 15
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
participants
  Maximum PR interval >=300 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum QRS Complex >=140 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum QTCF interval 450 to <480 msec | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Maximum QTCF interval 480 to <500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum QTCF interval >=500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR interval increase from baseline >=25/50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS complex increase from baseline >=50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTCF interval increase from baseline 30 to 60 msec | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  QTCF interval increase from baseline >=60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Hypoglycemic Adverse Event Based on Capillary Glucose Levels
Description: Capillary blood glucose levels were collected to observe any hypoglycemic adverse events. Hypoglycemia was assessed as following categories; Severe hypoglycemia (1. Participant was unable to treat himself/herself, requiring assistance of another person to actively administer carbohydrate, glucagon 2. Exhibited one of following neurological symptoms memory loss, uncontrollable behavior, irrational behavior, unusual difficulty in awakening, suspected seizure, seizure or loss of consciousness, 3. Glucose <50 mg/dL confirmed on repeat measure); Documented symptomatic hypoglycemia (1. Symptoms of hypoglycaemia accompanied by a measured glucose concentration <=70 mg/dL); asymptomatic hypoglycemia (not accompanied by typical symptoms of hypoglycaemia but with a measured glucose concentration <=70 mg/dL), and probable hypoglycemia (typical symptoms of hypoglycaemia are not accompanied by a glucose determination, but was presumably caused by a plasma glucose concentration <=70 mg/dL).
Time Frame: Day 0 up to Day 22
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
participants
  Severe Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Documented Symptomatic Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asymptomatic Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Probable Symptomatic Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Blood Glucose Abnormalities
Description: Criteria for blood glucose abnormality: Blood glucose levels <0.6*lower limit of normal (LLN) or >1.5*upper limit of normal (ULN).
Time Frame: Day -1 up to Day 15
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
participants
  <0.6*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >1.5*ULN | 7 | 6 | 6 | 6 | 6 | 5 | 3 | 9

8. Primary Outcome: Number of Participants With Anti-Drug Antibodies (ADA): Day 1
Description: Assays for the determination of human anti-drug (Anti-PF-05231023) antibodies (ADA) was performed.
Time Frame: Day 1
Population: Safety population included all participants who received at least 1 dose of study medication. No participant in the placebo group was assessed for this time point of outcome measure, hence results were not reported for the same.
Measure: Number; unit: participants
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10
participants | 0 | 1 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Anti-Drug Antibodies (ADA): Day 8
Description: Assays for the determination of human anti-drug (Anti-PF-05231023) antibodies (ADA) was performed.
Time Frame: Day 8
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Anti-Drug Antibodies (ADA): Day 15
Description: Assays for the determination of human anti-drug (Anti-PF-05231023) antibodies (ADA) was performed.
Time Frame: Day 15
Population: Safety population included all participants who received at least 1 dose of study medication. No participant in the placebo group was assessed for this time point of outcome measure, hence results were not reported for the same. 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg
Number analyzed (Participants) | 10 | 10 | 9 | 10 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Anti-Drug Antibodies (ADA): Day 22
Description: Assays for the determination of human anti-drug (Anti-PF-05231023) antibodies (ADA) was performed.
Time Frame: Day 22
Population: Safety population included all participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 9 | 9 | 1
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Anti-Drug Antibodies (ADA): Day 34
Description: Assays for the determination of human anti-drug (Anti-PF-05231023) antibodies (ADA) was performed.
Time Frame: Day 34
Population: Safety population. No participant was involved in groups: PF-05231023 0.5,1.5,5,15,50,100 mg and placebo for this time point of outcome measure, hence results were not reported for the same.'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | PF-05231023 200 mg
Number analyzed (Participants) | 1
participants | 0

13. Primary Outcome: Insulin-like Growth Factor - 1 (IGF-1), Insulin-like Growth Factor Binding Protein-1 (IGFBP-1), Insulin-like Growth Factor Binding Protein-2 (IGFBP-2), Growth Hormone (GH) Levels: Day 1
Description: Plasma samples for IGF-1, and GH were analyzed using a validated, sensitive, and specific immunochromatographic membrane assay (ICMA) fluorescence method. Plasma samples for IGFBP-1, IGFBP-2 were assayed using a validated, sensitive, and specific colorimetric sandwich (enzyme-linked immunosorbent assay) ELISA method.
Time Frame: Day 1
Population: Pharmacodynamic analysis set included all participants treated with PF-05231023 or placebo who had at least 1 pharmacodynamic endpoint. 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 5 | 10 | 9 | 12
nanogram per milliliter (ng/mL)
  IGF-1 | 137.2 (69.33) | 142.3 (47.10) | 143.4 (42.80) | 146.8 (50.97) | 128.4 (35.44) | 135.7 (59.12) | 153.1 (51.57) | 131.3 (34.71)
  IGFBP-1 | 1.83 (1.414) | 1.02 (0.525) | 2.63 (2.954) | 2.81 (2.454) | 1.20 (0.995) | 2.23 (3.138) | 2.88 (1.724) | 1.69 (1.292)
  IGFBP-2 | 173.5 (109.33) | 134.2 (50.00) | 143.8 (48.44) | 197.1 (147.01) | 108.8 (39.77) | 147.9 (89.58) | 204.7 (122.70) | 146.7 (79.50)
  GH | 0.178 (0.2981) | 0.121 (0.1521) | 0.133 (0.1629) | 0.222 (0.2189) | 0.316 (0.4162) | 0.296 (0.5557) | 0.448 (0.5928) | 0.079 (0.0355)

14. Primary Outcome: Insulin-like Growth Factor - 1 (IGF-1), Insulin-like Growth Factor Binding Protein-1 (IGFBP-1), Insulin-like Growth Factor Binding Protein-2 (IGFBP-2), Growth Hormone (GH) Levels: Day 2
Description: Plasma samples for IGF-1, and GH were analyzed using a validated, sensitive, and specific immunochromatographic membrane assay (ICMA) fluorescence method. Plasma samples for IGFBP-1, IGFBP-2 were assayed using a validated, sensitive, and specific colorimetric sandwich ELISA method.
Time Frame: Day 2
Population: Pharmacodynamic analysis set included all participants treated with PF-05231023 or placebo who had at least 1 pharmacodynamic endpoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
ng/mL
  IGF-1 | 141.1 (75.35) | 148.0 (47.00) | 163.5 (50.79) | 152.9 (51.08) | 145.0 (63.28) | 154.9 (55.30) | 168.4 (58.24) | 135.7 (33.89)
  IGFBP-1 | 2.72 (2.068) | 2.68 (1.570) | 2.37 (2.489) | 4.37 (4.093) | 2.67 (1.830) | 2.41 (1.711) | 4.49 (2.824) | 3.01 (2.954)
  IGFBP-2 | 153.1 (80.23) | 130.2 (43.42) | 154.4 (47.72) | 200.7 (171.17) | 117.7 (41.88) | 174.1 (104.64) | 212.6 (137.72) | 160.1 (87.53)
  GH | 0.230 (0.3135) | 0.369 (0.7146) | 0.182 (0.2109) | 0.386 (0.3823) | 0.316 (0.3116) | 0.407 (0.4363) | 0.620 (0.4641) | 0.498 (0.8284)

15. Primary Outcome: Insulin-like Growth Factor - 1 (IGF-1), Insulin-like Growth Factor Binding Protein-1 (IGFBP-1), Insulin-like Growth Factor Binding Protein-2 (IGFBP-2), Growth Hormone (GH) Levels: Day 3
Description: as for outcome 14
Time Frame: Day 3
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: nanogram per millileter (ng/mL)
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
nanogram per millileter (ng/mL)
  IGF-1 | 140.1 (62.82) | 147.5 (45.10) | 158.6 (46.26) | 164.2 (57.90) | 156.3 (75.73) | 149.8 (57.41) | 178.5 (53.85) | 137.7 (33.10)
  IGFBP-1 | 2.30 (1.910) | 2.57 (1.947) | 2.38 (2.863) | 3.00 (2.682) | 4.27 (4.803) | 2.70 (3.519) | 3.10 (1.694) | 2.00 (1.393)
  IGFBP-2 | 160.4 (106.14) | 135.7 (47.46) | 144.4 (43.00) | 188.2 (138.45) | 129.1 (42.61) | 155.0 (99.66) | 223.3 (120.05) | 145.2 (61.69)
  GH | 0.186 (0.2030) | 0.192 (0.1165) | 0.273 (0.3549) | 0.312 (0.3008) | 0.432 (0.6493) | 0.406 (0.3544) | 0.588 (0.4084) | 0.169 (0.1647)

16. Primary Outcome: Insulin-like Growth Factor - 1 (IGF-1), Insulin-like Growth Factor Binding Protein-1 (IGFBP-1), Insulin-like Growth Factor Binding Protein-2 (IGFBP-2), Growth Hormone (GH) Levels: Day 5
Description: as for outcome 14
Time Frame: Day 5
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: nanogram per millileter (ng/mL)
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
nanogram per millileter (ng/mL)
  IGF-1 | 138.4 (74.86) | 156.1 (40.03) | 152.7 (48.18) | 155.4 (54.29) | 136.9 (54.82) | 143.6 (54.03) | 163.6 (44.96) | 137.0 (27.00)
  IGFBP-1 | 2.45 (2.186) | 2.36 (1.629) | 2.61 (2.497) | 2.93 (2.547) | 4.02 (4.484) | 2.64 (3.102) | 3.11 (1.805) | 2.31 (2.466)
  IGFBP-2 | 169.1 (101.02) | 129.4 (44.14) | 152.4 (61.19) | 193.1 (137.11) | 135.5 (43.32) | 156.1 (117.61) | 207.9 (97.73) | 150.1 (69.66)
  GH | 0.190 (0.2492) | 0.146 (0.0802) | 0.169 (0.1788) | 0.233 (0.1884) | 0.271 (0.3159) | 0.188 (0.1641) | 0.484 (0.4962) | 0.216 (0.2418)

17. Primary Outcome: Insulin-like Growth Factor - 1 (IGF-1), Insulin-like Growth Factor Binding Protein-1 (IGFBP-1), Insulin-like Growth Factor Binding Protein-2 (IGFBP-2), Growth Hormone (GH) Levels: Day 7
Description: as for outcome 14
Time Frame: Day 7
Population: Pharmacodynamic analysis set included all participants treated with PF-05231023 or placebo who had at least 1 pharmacodynamic endpoint. Here,'n' signifies participants who were evaluable at each specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
nanogram per milliliter (ng/mL)
  IGF-1 (n=10,10,10,10,10,10,10,14) | 142.1 (73.55) | 151.0 (47.72) | 152.3 (54.13) | 157.1 (61.32) | 130.4 (55.44) | 143.9 (59.06) | 154.1 (41.88) | 132.5 (28.07)
  IGFBP-1 (n=10,10,10,10,10,9,10,14) | 4.67 (3.533) | 2.77 (2.113) | 3.03 (3.261) | 2.98 (3.948) | 2.61 (2.348) | 2.80 (3.440) | 3.39 (1.824) | 3.46 (4.404)
  IGFBP-2 (n=10,10,10,10,10,9,10,14) | 187.7 (107.34) | 116.5 (30.62) | 166.4 (48.32) | 178.7 (126.83) | 132.8 (46.18) | 173.8 (148.78) | 229.8 (118.94) | 154.7 (88.03)
  GH (n=10,10,10,10,10,10,10,14) | 0.233 (0.2506) | 0.112 (0.0738) | 0.108 (0.0760) | 0.254 (0.3971) | 0.142 (0.1003) | 0.120 (0.1067) | 0.320 (0.1942) | 0.201 (0.2193)

18. Primary Outcome: Insulin-like Growth Factor - 1 (IGF-1), Insulin-like Growth Factor Binding Protein-1 (IGFBP-1), Insulin-like Growth Factor Binding Protein-2 (IGFBP-2), Growth Hormone (GH) Levels: Day 15
Description: as for outcome 14
Time Frame: Day 15
Population: Pharmacodynamic analysis set included all participants treated with PF-05231023 or placebo who had at least 1 pharmacodynamic endpoint. 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure. 'n' signifies participants who were evaluable for each specified parameter for each arm, respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 10 | 10 | 9 | 9 | 14
nanogram per milliliter (ng/mL)
  IGF-1 (n=10,10,9,10,10,9,9,14) | 117.7 (55.26) | 132.6 (42.72) | 116.7 (38.99) | 131.2 (45.53) | 106.2 (44.50) | 123.2 (51.08) | 126.3 (40.32) | 112.5 (25.85)
  IGFBP-1 (n=10,10,9,10,10,9,9,14) | 3.30 (1.999) | 2.59 (1.573) | 2.90 (3.357) | 2.28 (2.262) | 2.70 (2.186) | 3.23 (3.567) | 3.36 (2.261) | 2.11 (1.690)
  IGFBP-2 (n=10,10,9,10,10,9,9,14) | 215.6 (89.55) | 154.7 (38.39) | 157.3 (60.35) | 240.8 (177.76) | 155.4 (49.16) | 193.1 (145.98) | 247.3 (145.61) | 181.6 (129.74)
  GH (n=10,10,9,10,10,9,9,14) | 0.216 (0.2557) | 0.135 (0.1039) | 0.133 (0.1111) | 0.115 (0.0920) | 0.090 (0.0927) | 0.161 (0.1388) | 0.183 (0.2236) | 0.180 (0.1628)

19. Primary Outcome: Insulin-like Growth Factor Binding Protein-3 (IGFBP-3) Levels: Day 1
Description: Plasma samples were assayed using a validated, sensitive, and specific ICMA fluorescence method.
Time Frame: Day 1
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 5 | 10 | 9 | 12
microgram per milliliter (mcg/mL) | 3.09 (1.028) | 4.03 (1.325) | 3.80 (1.026) | 3.47 (0.804) | 3.52 (1.260) | 3.44 (1.198) | 3.52 (1.003) | 3.66 (0.925)

20. Primary Outcome: Insulin-like Growth Factor Binding Protein-3 (IGFBP-3) Levels: Day 2
Description: Plasma samples were assayed using a validated, sensitive, and specific ICMA fluorescence method.
Time Frame: Day 2
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
mcg/mL | 3.11 (0.983) | 4.04 (1.211) | 3.78 (0.887) | 3.49 (0.839) | 3.79 (1.440) | 3.53 (1.069) | 3.53 (0.888) | 3.63 (0.986)

21. Primary Outcome: Insulin-like Growth Factor Binding Protein-3 (IGFBP-3) Levels: Day 3
Description: Plasma samples were assayed using a validated, sensitive, and specific ICMA fluorescence method.
Time Frame: Day 3
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
mcg/mL | 3.14 (0.964) | 3.99 (1.180) | 3.82 (0.957) | 3.56 (0.957) | 3.69 (1.433) | 3.38 (0.907) | 3.54 (0.948) | 3.75 (0.924)

22. Primary Outcome: Insulin-like Growth Factor Binding Protein-3 (IGFBP-3) Levels: Day 5
Description: Plasma samples were assayed using a validated, sensitive, and specific ICMA fluorescence method.
Time Frame: Day 5
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
mcg/mL | 3.12 (0.930) | 3.98 (1.269) | 3.89 (1.026) | 3.53 (0.830) | 3.41 (1.242) | 3.27 (1.024) | 3.32 (0.747) | 3.60 (0.969)

23. Primary Outcome: Insulin-like Growth Factor Binding Protein-3 (IGFBP-3) Levels: Day 7
Description: Plasma samples were assayed using a validated, sensitive, and specific ICMA fluorescence method.
Time Frame: Day 7
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 14
mcg/mL | 3.27 (1.049) | 4.01 (1.297) | 3.84 (0.969) | 3.58 (0.968) | 3.43 (1.378) | 3.25 (0.996) | 3.32 (0.721) | 3.51 (0.901)

24. Primary Outcome: Insulin-like Growth Factor Binding Protein-3 (IGFBP-3) Levels: Day 15
Description: Plasma samples were assayed using a validated, sensitive, and specific ICMA fluorescence method.
Time Frame: Day 15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 10 | 10 | 9 | 9 | 14
mcg/mL | 2.88 (0.884) | 3.72 (1.166) | 3.51 (0.961) | 3.25 (0.654) | 3.11 (1.135) | 3.30 (0.890) | 3.20 (0.876) | 3.46 (0.920)

25. Primary Outcome: Number of Participants With Abnormal Cardiac Rhythms Recorded by Telemetry
Description: Criteria for abnormal cardiac rhythms was based on investigator's discretion and were reported as adverse event (AE), as planned.
Time Frame: From 2 hours (H) pre-dose for intravenous bolus or 2 H prior to the start of infusion on Day 1 up to 8 H post-dose for bolus or 8 H following the end of the infusion on Day 1
Population: Data was not collected since this outcome measure was not analyzed as per Sponsor's discretion.
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Area Under the Curve From Time Zero to Time of Last Quantifiable Plasma Concentration (AUClast) of PF-05231023
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
  Participants who received PF-05231023 with C-terminal and N-terminal AUClast were reported.
Time Frame: Hour(H)-1(prior to start of infusion[In] or 1 H pre-dose to bolus[Bo]),H-0.5(0.5 H post start of In or 0.5 H pre-dose to Bo),H 0(end of In or prior to Bo),0.25,0.5,1,1.5,2,3,5,8,12 H post end of In or post-dose to Bo on Day 1;Day 2,3,4,5,6,8,15,22
Population: Pharmacokinetic (PK) parameter analysis set included all participants randomized and treated who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Standard Deviation); unit: ng*hour[H]/mL
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10
ng*hour[H]/mL
  C-terminal | 672.3 (364.50) | 2573 (475.73) | 10220 (4059.2) | 29390 (6697.4) | 95120 (13749) | 244200 (83895) | 409300 (135030)
  N-terminal | 2957 (1887.2) | 11630 (4363.6) | 47650 (10833) | 168600 (50175) | 564600 (161560) | 121100 (386970) | 280000 (756220)

27. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-05231023
Description: Participants who received PF-05231023 with C-terminal and N-terminal Tmax were reported.
Time Frame: as for outcome 26
Population: PK parameter analysis set included all participants randomized and treated who had at least 1 of the PK parameters of primary interest.
Measure: Median (Full Range); unit: hour
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10
hour
  C-terminal | 0.250 [0.250 to 0.533] | 0.250 [0.250 to 0.500] | 1.50 [1.50 to 3.00] | 1.50 [1.02 to 2.53] | 1.26 [1.00 to 1.50] | 1.50 [1.00 to 6.00] | 1.02 [1.00 to 2.50]
  N-terminal | 0.250 [0.250 to 3.03] | 0.250 [0.250 to 1.00] | 1.50 [1.50 to 6.00] | 1.50 [1.02 to 2.50] | 1.26 [1.00 to 6.00] | 1.50 [1.00 to 2.50] | 1.50 [1.00 to 2.52]

28. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-05231023
Description: Participants who received PF-05231023 with C-terminal and N-terminal Cmax were reported.
Time Frame: as for outcome 26
Population: as for outcome 27
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10
ng/mL
  C-terminal | 110.7 (40.994) | 347.9 (61.165) | 1360 (1264.9) | 3324 (656.74) | 11730 (4857.6) | 28740 (8031.1) | 47780 (13784)
  N-terminal | 121.0 (44.923) | 393.2 (75.603) | 1199 (386.56) | 3693 (714.42) | 14180 (3928.7) | 28850 (6375.5) | 61910 (8125.5)

29. Secondary Outcome: Plasma Terminal Half-Life (t1/2) of PF-05231023
Description: Plasma terminal half-life is the time measured for the plasma concentration to decrease by one half at the terminal phase. Participants who received PF-05231023 with C-terminal and N-terminal t1/2 were reported.
Time Frame: as for outcome 26
Population: PK parameter analysis set included all participants randomized and treated who had at least 1 of the PK parameters of primary interest. 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.'n' signifies participants who were evaluable for each specified parameter for each arm, respectively.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg
Number analyzed (Participants) | 7 | 10 | 10 | 9 | 10 | 10 | 10
hour
  C-terminal (n=2,10,10,9,10,10,10) | NA (NA) — Data was not reported since less than 3 participants were evaluable. | 6.504 (1.0814) | 7.168 (1.2433) | 7.143 (1.5009) | 7.748 (1.1304) | 7.502 (0.9999) | 7.302 (1.7117)
  N-terminal (n=7,9,10,10,9,10,10) | 31.49 (6.5685) | 37.64 (9.0438) | 66.54 (12.792) | 77.39 (11.979) | 81.52 (12.599) | 87.69 (16.556) | 96.64 (8.0925)

30. Secondary Outcome: Apparent Clearance (CL) of PF-05231023 for Intravenous Bolus Dosing
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.Participants who received PF-05231023 with C-terminal and N-terminal CL were reported.
Time Frame: Hour (H)-1 (1 H pre-dose to bolus [Bo]),H-0.5(0.5 H pre-dose to Bo),H 0 (prior to Bo),0.25,0.5,1,1.5,2,3,5,8,12 H post-dose to Bo on Day 1;Day 2,3,4,5,6,8,15,22
Population: PK parameter analysis set included all participants randomized and treated who had at least 1 of the PK parameters of primary interest. 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure. 'n' signifies participants who were evaluable for each specified parameter for each arm, respectively.
Measure: Geometric Mean (Standard Deviation); unit: liter per hour
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg
Number analyzed (Participants) | 7 | 10 | 10 | 9 | 10 | 10 | 10
liter per hour
  C-terminal (n=2,10,10,9,10,10,10) | NA (NA) — Data was not reported since less than 3 participants were evaluable. | 0.5368 (0.0972) | 0.4642 (0.15736) | 0.4974 (0.12295) | 0.5245 (0.0892) | 0.4092 (0.12015) | 0.4883 (0.25652)
  N-terminal (n=7,9,10,10,9,10,10) | 0.1057 (0.0459) | 0.1282 (0.0417) | 0.1014 (0.0203) | 0.0879 (0.03216) | 0.08611 (0.02916) | 0.08050 (0.0256) | 0.07021 (0.0186)

31. Secondary Outcome: Apparent Volume of Distribution (Vz) of PF-05231023
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. PF-05231023 with C-terminal and N-terminal Vz were reported.
Time Frame: as for outcome 26
Population: as for outcome 30
Measure: Geometric Mean (Standard Deviation); unit: Liter
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg
Number analyzed (Participants) | 7 | 10 | 10 | 9 | 10 | 10 | 10
Liter
  C-terminal (n=2,10,10,9,10,10,10 ) | NA (NA) — Data was not reported since less than 3 participants were evaluable. | 4.977 (0.93206) | 4.741 (1.1834) | 5.029 (0.81502) | 5.799 (1.5559) | 4.397 (1.1511) | 5.014 (1.2498)
  N-terminal (n=7,9,10,10,9,10,10) | 4.709 (0.82966) | 6.758 (1.1934) | 9.526 (2.2753) | 9.704 (2.1259) | 10.01 (2.9519) | 9.979 (2.7792) | 9.767 (2.5208)

32. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of PF-05231023
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞). PF-05231023 with C-terminal and N-terminal AUC (0 - ∞) were reported.
Time Frame: as for outcome 26
Population: PK parameter analysis set included all participants randomized and treated who have at least 1 of the PK parameters of primary interest. 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure. 'n' signifies participants who were evaluable for each specified parameter for each arm, respectively.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg
Number analyzed (Participants) | 7 | 10 | 10 | 9 | 10 | 10 | 10
ng*hr/ml
  C-terminal (n=2,10,10,9,10,10,10) | NA (NA) — Data was not reported since less than 3 participants were evaluable. | 2793 (557.86) | 10770 (3999.8) | 30140 (7079.3) | 95350 (13817) | 244300 (84238) | 409700 (135300)
  N-terminal (n=7,9,10,10,9,10,10) | 4726 (1594.5) | 11700 (4305.5) | 49340 (10835) | 170600 (50735) | 581000 (168820) | 1241000 (395290) | 2848000 (779810)

33. Secondary Outcome: Back-extrapolated Concentration at Time Zero (C0) of PF-05231023
Description: C0 was estimated by back-extrapolating from the first 2 concentration values using the log-linear regression on the first 2 data points (where second concentration was less than [<] first concentration) to back-extrapolate C0. PF-05231023 with C-terminal and N-terminal C0 were reported.
Time Frame: 0.25 H post-dose to Bo on Day 1
Population: PK parameter analysis set included all participants randomized and treated who have at least 1 of the PK parameters of primary interest. C0 was calculated for cohort 1 (group: PF-05231023 0.5 mg) and 2 (group: PF-05231023 1.5 mg) only as per planned analysis, hence results for the same reported.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg
Number analyzed (Participants) | 10 | 10
ng/mL
  C-terminal | 116.7 (47.581) | 363.0 (81.903)
  N-terminal | 131.8 (47.543) | 415.4 (81.456)

34. Secondary Outcome: Volume of Distribution at Steady State (Vss) of PF-05231023
Description: Vss was calculated by dividing the area under the first moment curve from time zero to infinity [AUMC(0-∞)] with the product of area under the curve from time zero to extrapolated infinite time [AUC (0 - ∞)] and apparent clearance (CL). PF-05231023 with C-terminal and N-terminal Vss were reported.
Time Frame: as for outcome 26
Population: as for outcome 32
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg
Number analyzed (Participants) | 7 | 10 | 10 | 9 | 10 | 10 | 10
L
  C-terminal (n=2,10,10,9,10,10,10) | NA (NA) — Data was not reported since less than 3 participants were evaluable. | 4.897 (0.9277) | 4.596 (1.2589) | 5.023 (0.96722) | 5.650 (1.9178) | 4.082 (1.1896) | 4.655 (1.0748)
  N-terminal (n=7,9,10,10,9,10,10) | 4.544 (0.81713) | 6.151 (1.1762) | 7.165 (1.4032) | 7.322 (1.2447) | 7.022 (1.4714) | 7.004 (1.4774) | 7.197 (1.4347)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-05231023 0.5 mg | PF-05231023 1.5 mg | PF-05231023 5 mg | PF-05231023 15 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 200 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/14
Other Adverse Events (participants affected / at risk) | 4/10 | 3/10 | 3/10 | 2/10 | 7/10 | 2/10 | 8/10 | 5/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05231023 0.5 mg (N=10) | PF-05231023 1.5 mg (N=10) | PF-05231023 5 mg (N=10) | PF-05231023 15 mg (N=10) | PF-05231023 50 mg (N=10) | PF-05231023 100 mg (N=10) | PF-05231023 200 mg (N=10) | Placebo (N=14)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 6 | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Administration site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Results for C0 and Vss was included as secondary endpoints as per change in the planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.